CLINICAL TRIAL: NCT05985044
Title: Living With Multimorbidity: Symptom Management Across the Illness Trajectory
Brief Title: Living With Multimorbidity: CO-ORDINATE Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00244792; P30NR018093 (NIH)
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Multimorbidity; Quality of Life; Symptom Management
MeSH Terms: interventions — Palliative Care; Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): A patient-centered Care cO-ORDInatioN And sympTom managEment (CO-ORDINATE) intervention
  Interventions: Other: Care cO-ORDInatioN And sympTom managEment (CO-ORDINATE) Intervention

INTERVENTIONS:
Other: Care cO-ORDInatioN And sympTom managEment (CO-ORDINATE) Intervention — The intervention consists of the following four components: i) needs assessment; ii) question prompt list; iii) goals discussion and; iv) symptom assessment and tracking. The intervention will start with the enrolment of a patient living with multimorbidity. The intervention consists of one in-person pre-discharge visit by the study team and four follow-up telephone calls (at 48 hours, 1 week, 4 weeks, and 6 weeks post-discharge).

SUMMARY:
Multimorbidity is common and is the coexistence of two or more chronic conditions in the same individual. People with multimorbidity suffer from a high symptom burden, directly affecting quality of life (QOL). Hospitalization can be a window of opportunity to initiate interventions to promote recovery and resilience and enhance QOL. However, interventions targeting the symptom trajectory and burden of patients with multimorbidity are lacking. Thus, the investigators envisage a nurse-led pre-discharge intervention augmented by telephone support, focusing on care coordination and symptom management. This approach is anticipated to help reduce symptom burden and improve QOL.

DETAILED DESCRIPTION:
Aim 1: Describe the symptom trajectory and burden from the perspectives of patients, family caregivers, and health professionals and collectively develop a symptom management toolkit; and

Aim 2: Refine and pilot test the nurse-driven symptom management toolkit/intervention to decrease the symptom burden and increase the QOL of critically ill adults with multimorbidity.

Interventional study (Aim 2):

The study aims to test the feasibility of the Care cOORDInatioN and sympTom managEment (COORDINATE) intervention developed from Aim 1 using an experienced-based co-design methodology. A single-arm feasibility study will be implemented with assumptions on the effectiveness of the COORDINATE intervention on outcomes such as symptom burden and quality of life will be evaluated.

Sample and Setting:

Individuals aged 55 years and older, living with two or more chronic health conditions, and willing to provide informed consent will be included in the study. The exclusion criteria include if participants cannot speak English or have a documented cognitive impairment that would prevent participation. Patients will be approached in the Intermediate Care Unit (IMCU) of an academic teaching hospital while the participants are in-patient before discharge.

Intervention Components and Timing:

The intervention consists of four components- i) needs assessment; ii) question prompt list; iii) goals discussion and; iv) symptom assessment and tracking. The intervention will start with the enrolment of a patient living with multimorbidity. The intervention consists of one in-person pre-discharge visit by the study team and four follow-up telephone calls (at 48 hours, 1 week, 4 weeks, and 6 weeks post-discharge).

Primary Outcomes

1. Symptom Burden
2. Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* English speakers who are planned for discharge from Johns Hopkins Hospital (JHH) IMCU
* Who meet the criteria for being admitted to IMCU and planned discharge with multimorbidity as defined by two or more chronic conditions.

Exclusion Criteria:

* Who can not provide informed consent or have documented cognitive impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binu Koirala, PhD, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Koirala B, Badawi S, Frost S, Ferguson C, Hager DN, Street L, Perrin N, Dennison Himmelfarb C, Davidson P. Study protocol for Care cOORDInatioN And sympTom managEment (COORDINATE) programme: a feasibility study. BMJ Open. 2023 Dec 18;13(12):e072846. doi: 10.1136/bmjopen-2023-072846. PMID 38110376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participant was approached and recruited in the Intermediate Care Unit (IMCU) of an academic teaching hospital while the participants are in-patient before discharge. The recruitment of eligible participant took approximately 9 months from November 16, 2022 to August 2, 2023.
Pre-assignment Details: Out of the 27 participants who signed the informed consent, 25 completed the baseline survey and received the intervention. Two participants did not complete the baseline data collection and could not be reached after signing the consent form.
Groups:
- Intervention: The participants received the Care cO-ORDInatioN And sympTom managEment (CO-ORDINATE) intervention, which includes the following four components: i) needs assessment, ii) question prompt list, iii) goals discussion, and iv) symptom assessment and tracking. The intervention comprises one in-person pre-discharge visit by the study team and four follow-up telephone calls conducted at 48 hours, 1 week, 4 weeks, and 6 weeks post-discharge.
Period: Overall Study
Arm/Group | Intervention
Started | 25 (25 completed baseline data collection.)
Completed | 10 (10 completed self-reported surveys at 3 months' follow-up.)
Not Completed | 15
Not completed — Death | 6
Not completed — Lost to Follow-up | 4
Not completed — Incapacitation | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Symptom burden - Pain [Mean (Standard Deviation); unit: units on a scale] — The Symptom burden assessed by Edmonton Symptom Assessment System (ESAS) score; with ratings ranging from 0 (none, best) to 10 (worst). Mean of participant choice is reported.
  units on a scale | 4.34 (3.63)
Symptom burden - Tiredness [Mean (Standard Deviation); unit: units on a scale] — The Symptom burden assessed by Edmonton Symptom Assessment System (ESAS) score; with ratings ranging from 0 (none, best) to 10 (worst). Mean of participant choice is reported.
  units on a scale | 3.64 (2.89)
Symptom burden - Drowsiness [Mean (Standard Deviation); unit: units on a scale] — The Symptom burden assessed by Edmonton Symptom Assessment System (ESAS) score; with ratings ranging from 0 (none, best) to 10 (worst). Mean of participant choice is reported.
  units on a scale | 2.48 (2.76)
Symptom burden - Nausea [Mean (Standard Deviation); unit: units on a scale] — The Symptom burden assessed by Edmonton Symptom Assessment System (ESAS) score; with ratings ranging from 0 (none, best) to 10 (worst). Mean of participant choice is reported.
  units on a scale | 1.52 (2.87)
Symptom burden - Lack of appetite [Mean (Standard Deviation); unit: units on a scale] — The Symptom burden assessed by Edmonton Symptom Assessment System (ESAS) score; with ratings ranging from 0 (none, best) to 10 (worst). Mean of participant choice is reported.
  units on a scale | 1.02 (2.19)
Symptom burden - Shortness of breath [Mean (Standard Deviation); unit: units on a scale] — The Symptom burden assessed by Edmonton Symptom Assessment System (ESAS) score; with ratings ranging from 0 (none, best) to 10 (worst). Mean of participant choice is reported.
  units on a scale | 2.16 (2.76)
Symptom burden - Depression [Mean (Standard Deviation); unit: units on a scale] — The Symptom burden assessed by Edmonton Symptom Assessment System (ESAS) score; with ratings ranging from 0 (none, best) to 10 (worst). Mean of participant choice is reported.
  units on a scale | 1.78 (3.19)
Symptom burden - Anxiety [Mean (Standard Deviation); unit: units on a scale] — The Symptom burden assessed by Edmonton Symptom Assessment System (ESAS) score; with ratings ranging from 0 (none, best) to 10 (worst). Mean of participant choice is reported.
  units on a scale | 2.3 (2.97)
Symptom burden - Well-being [Mean (Standard Deviation); unit: units on a scale] — The Symptom burden assessed by Edmonton Symptom Assessment System (ESAS) score; with ratings ranging from 0 (none, best) to 10 (worst). Mean of participant choice is reported.
  units on a scale | 4.48 (3.27)
Quality of Life - Physical functioning [Mean (Standard Deviation); unit: units on a scale] — Quality of Life assessed by Short Form Survey (SF-36) score; score range 0 to 100. Higher score is better quality of life.
  units on a scale | 43.33 (30.31)
Quality of Life - Role Physical [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life assessed by Short Form Survey (SF-36) score; score range 0 to 100. Higher score is better quality of life.
  units on a scale | 27.08 (36.05)
Quality of Life -Role Emotional [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life assessed by Short Form Survey (SF-36) score; score range 0 to 100. Higher score is better quality of life.
  units on a scale | 48.61 (46.08)
Quality of Life - Vitality [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life assessed by Short Form Survey (SF-36) score; score range 0 to 100. Higher score is better quality of life.
  units on a scale | 42.08 (22.89)
Quality of Life - Mental Health [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life assessed by Short Form Survey (SF-36) score; score range 0 to 100. Higher score is better quality of life.
  units on a scale | 65 (26.49)
Quality of Life - Social Functioning [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life assessed by Short Form Survey (SF-36) score; score range 0 to 100. Higher score is better quality of life.
  units on a scale | 51.04 (35.72)
Quality of Life - Social Functioning [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life assessed by Short Form Survey (SF-36) score; score range 0 to 100. Higher score is better quality of life.
  units on a scale | 51.04 (35.72)
Quality of Life - General health [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life assessed by Short Form Survey (SF-36) score; score range 0 to 100. Higher score is better quality of life.
  units on a scale | 49.58 (22.07)

OUTCOME MEASURES:

1. Primary Outcome: Symptom Burden Assessed by Edmonton Symptom Assessment System (ESAS) Score - Pain
Description: The ESAS questionnaire is used to rate the intensity of common symptoms including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath; with ratings ranging from 0 (none, best) to 10 (worst).
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
score on a scale
  Baseline | 5 [0 to 8]
  6-week: number analyzed (Participants) | 7
  6-week | 4 [1 to 6]
  3-month: number analyzed (Participants) | 10
  3-month | 5 [2 to 7]

2. Primary Outcome: Symptom Burden Assessed by Edmonton Symptom Assessment System (ESAS) Score - Tiredness
Description: as for outcome 1
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
score on a scale
  Baseline | 3 [2 to 5]
  6-week: number analyzed (Participants) | 7
  6-week | 3 [3 to 4]
  3-month: number analyzed (Participants) | 10
  3-month | 6 [3 to 7]

3. Primary Outcome: Symptom Burden Assessed by Edmonton Symptom Assessment System (ESAS) Score - Drowsiness
Description: as for outcome 1
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
score on a scale
  Baseline | 2 [0 to 5]
  6-week: number analyzed (Participants) | 7
  6-week | 3 [0 to 4]
  3-month: number analyzed (Participants) | 10
  3-month | 5 [2 to 6]

4. Primary Outcome: Symptom Burden Assessed by Edmonton Symptom Assessment System (ESAS) Score - Nausea
Description: as for outcome 1
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
score on a scale
  Baseline | 0 [0 to 0]
  6-week: number analyzed (Participants) | 7
  6-week | 0 [0 to 0.3]
  3-month: number analyzed (Participants) | 10
  3-month | 1 [0 to 2.5]

5. Primary Outcome: Symptom Burden Assessed by Edmonton Symptom Assessment System (ESAS) Score - Lack of Appetite
Description: as for outcome 1
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
score on a scale
  Baseline | 0 [0 to 0]
  6-week: number analyzed (Participants) | 7
  6-week | 1 [0 to 6]
  3-month: number analyzed (Participants) | 10
  3-month | 3.3 [1 to 4]

6. Primary Outcome: Symptom Burden Assessed by Edmonton Symptom Assessment System (ESAS) Score - Shortness of Breath
Description: as for outcome 1
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
score on a scale
  Baseline | 0 [0 to 4]
  6-week: number analyzed (Participants) | 7
  6-week | 3 [1 to 4]
  3-month: number analyzed (Participants) | 10
  3-month | 5 [3 to 5]

7. Primary Outcome: Symptom Burden Assessed by Edmonton Symptom Assessment System (ESAS) Score - Depression
Description: as for outcome 1
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
score on a scale
  Baseline | 0 [0 to 3]
  6-week: number analyzed (Participants) | 7
  6-week | 3 [1 to 5]
  3-month: number analyzed (Participants) | 10
  3-month | 4.5 [1 to 6]

8. Primary Outcome: Symptom Burden Assessed by Edmonton Symptom Assessment System (ESAS) Score - Anxiety
Description: as for outcome 1
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
score on a scale
  Baseline | 0 [0 to 5]
  6-week: number analyzed (Participants) | 7
  6-week | 2 [0.5 to 6]
  3-month: number analyzed (Participants) | 10
  3-month | 2.5 [0 to 5]

9. Primary Outcome: Symptom Burden Assessed by Edmonton Symptom Assessment System (ESAS) Score - Well-being
Description: as for outcome 1
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
score on a scale
  Baseline | 5 [0 to 7]
  6-week: number analyzed (Participants) | 7
  6-week | 4 [3.3 to 6.5]
  3-month: number analyzed (Participants) | 10
  3-month | 3.3 [2 to 5]

10. Primary Outcome: Quality of Life Assessed by Short Form Survey (SF-36) Score - Physical Functioning
Description: Short Form Survey (SF-36) is a 36-item self-reported quality of life that covers 8 domains; score range 0 to 100. Higher score is better quality of life.
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 24
score on a scale
  Baseline | 50 [12.5 to 62.5]
  6-week: number analyzed (Participants) | 7
  6-week | 40 [25 to 60]
  3-month: number analyzed (Participants) | 10
  3-month | 32.5 [10 to 65]

11. Primary Outcome: Quality of Life Assessed by Short Form Survey (SF-36) Score - Role Physical
Description: as for outcome 10
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 24
score on a scale
  Baseline | 25 [0 to 25]
  6-week: number analyzed (Participants) | 7
  6-week | 0 [0 to 100]
  3-month: number analyzed (Participants) | 10
  3-month | 0 [0 to 75]

12. Primary Outcome: Quality of Life Assessed by Short Form Survey (SF-36) Score - Role Emotional
Description: as for outcome 10
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 24
score on a scale
  Baseline | 33.33 [0 to 100]
  6-week: number analyzed (Participants) | 7
  6-week | 33.33 [0 to 100]
  3-month: number analyzed (Participants) | 10
  3-month | 16.67 [0 to 100]

13. Primary Outcome: Quality of Life Assessed by Short Form Survey (SF-36) Score - Vitality
Description: as for outcome 10
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 24
score on a scale
  Baseline | 45 [22.5 to 60]
  6-week: number analyzed (Participants) | 7
  6-week | 50 [35 to 50]
  3-month: number analyzed (Participants) | 10
  3-month | 52.5 [50 to 65]

14. Primary Outcome: Quality of Life Assessed by Short Form Survey (SF-36) Score - Mental Health
Description: as for outcome 10
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who competed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 24
score on a scale
  Baseline | 68 [48 to 88]
  6-week: number analyzed (Participants) | 7
  6-week | 68 [46 to 92]
  3-month: number analyzed (Participants) | 10
  3-month | 76 [44 to 88]

15. Primary Outcome: Quality of Life Assessed by Short Form Survey (SF-36) Score - Social Functioning
Description: as for outcome 10
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who completed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 24
score on a scale
  Baseline | 50 [25 to 87.5]
  6-week: number analyzed (Participants) | 7
  6-week | 62.5 [25 to 75]
  3-month: number analyzed (Participants) | 10
  3-month | 50 [25 to 75]

16. Primary Outcome: Quality of Life Assessed by Short Form Survey (SF-36) Score - Bodily Pain
Description: as for outcome 10
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who completed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 24
score on a scale
  Baseline | 38.75 [10 to 67.5]
  6-week: number analyzed (Participants) | 7
  6-week | 57.5 [42.5 to 67.5]
  3-month: number analyzed (Participants) | 10
  3-month | 50 [45 to 60]

17. Primary Outcome: Quality of Life Assessed by Short Form Survey (SF-36) Score - General Health
Description: as for outcome 10
Time Frame: Baseline, 6-weeks post intervention, 3 months post intervention
Population: Participants who completed the survey at each time point are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 24
score on a scale
  Baseline | 50 [30 to 65]
  6-week: number analyzed (Participants) | 7
  6-week | 45 [25 to 80]
  3-month: number analyzed (Participants) | 10
  3-month | 40 [30 to 60]

18. Secondary Outcome: Health-care Utilization - Total Healthcare Utilization
Description: Health-care utilization data will be retrieved from electronic medical records. The study team is defining healthcare utilization by identifying no. of total healthcare utilization, hospitalizations, emergency visits, and critical care admissions. Higher the numbers higher the healthcare utilization.
Time Frame: 3 months before and after entering the program
Population: One outlier was excluded from the data.
Measure: Median (Inter-Quartile Range); unit: Care utilization events
Arm/Group | Intervention
Number analyzed (Participants) | 24
Care utilization events
  3 months before entering the program | 1 [1 to 2]
  3 months after entering the program | 1 [0 to 2]

19. Secondary Outcome: Health-care Utilization - Emergency Department (ED) Visit s
Description: as for outcome 18
Time Frame: 3 months before and after entering the program
Population: Participants who had data available are reported.
Measure: Median (Inter-Quartile Range); unit: Care utilization events
Arm/Group | Intervention
Number analyzed (Participants) | 24
Care utilization events
  3 months before entering the program | 1 [1 to 2]
  3 months after entering the program | 1 [0 to 1.5]

20. Secondary Outcome: Health-care Utilization - Hospitalization
Description: Health-care utilization data will be retrieved from electronic medical records. The study team is defining healthcare utilization by identifying no. of total healthcare utilization, hospitalizations, emergency visits, and critical care admissions.. Higher the numbers higher the healthcare utilization.
Time Frame: 3 months before and after entering the program
Population: Participants who had data available are reported.
Measure: Median (Inter-Quartile Range); unit: Care utilization events
Arm/Group | Intervention
Number analyzed (Participants) | 24
Care utilization events
  3 months before entering the program | 1 [1 to 1]
  3 months after entering the program | 0 [0 to 1]

21. Secondary Outcome: Health-care Utilization - Critical Care Admission
Description: as for outcome 18
Time Frame: 3 months before and after entering the program
Population: Participants who had data available are reported.
Measure: Median (Inter-Quartile Range); unit: Care utilization events
Arm/Group | Intervention
Number analyzed (Participants) | 24
Care utilization events
  3 months before entering the program | 1 [1 to 1]
  3 months after entering the program | 0 [0 to 0.5]

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 6/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
Because of the feasibility design, the study is not powered. Hence, changes in primary and secondary outcomes over time (i.e., baseline vs 6 weeks and 3 months) must be considered carefully.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT05985044/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT05985044/ICF_001.pdf